CLINICAL TRIAL: NCT04320914
Title: High Intensity Laser Therapy (Classes IV) and Ibuprofen Gel Phonophoresis for Treating Knee Osteoarthritis Among People Living in Hilly Terrain: A Randomized, Double Blind, Controlled Study
Brief Title: High Intensity Laser Therapy (Classes IV) and Ibuprofen Gel Phonophoresis for Treating Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Collaborators: Himachal Pradesh Council for Science Technology and Environment (HIMCOSTE) (Unknown)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/IEC/140E; U1111-1237-6893 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Osteo Arthritis Knee
Keywords: Knee osteoarthritis; Incline walking; degeneration; Ultrasound; laser therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity LASER Therapy group (HILT) (Experimental): Fourty patients with chronic KOA in HILT group will receive Class IV LASER therapy. A Class IV LASER emits power more than 500 mW .
  Interventions: Other: High Intensity LASER Therapy
- Ibuprofen gel phonophoresis (IGP) group (Active Comparator): Patients with chronic KOA in IGP group will administered with continuous ultrasound set at a frequency of 1 MHz and an intensity of 1 W/cm2 was applied on a circular basis
  Interventions: Other: Ibuprofen gel phonophoresis

INTERVENTIONS:
Other: High Intensity LASER Therapy — The total energy will be delivered to the patient during one session will be 1,250 J through three phases of treatment.
  1. Initial phase (710 and 810 mJ/cm2 for a total of 500 J)
  2. Intermediate phase (handpiece will be applied on the joint line just proximal to the medial and lateral tibial condyles with 25 J, a fluency of 610 mJ/cm2, and a time of 14 s for each point and a total of 250 J)
  3. Final phase (same as the initial phase (500 J) except that scanning will be slow manual scanning ) The application time for all three phases will be approximately 15 min with the total energy delivered to the patient during one session of 1,250 J Duration of the treatment will be 8 minutes in one session/knee joint for each day for 3 days/week for 8 weeks.
  Other Names: HILT
  Arms: High Intensity LASER Therapy group (HILT)
Other: Ibuprofen gel phonophoresis — Continuous ultrasound set at a frequency of 1 MHz and an intensity of 1 W/cm2 was applied on a circular basis. Each treatment session will last for 8 min with one session each day for 3 days/week for 8 weeks.
  Other Names: IGP
  Arms: Ibuprofen gel phonophoresis (IGP) group

SUMMARY:
A total of 80 patients with knee osteoarthritis (KOA) aged between fourty five and seventy years will be recruited by simple random sampling to participate in two group, randomized, double blind, controlled study. Recruited patients will be randomly divided in to two groups high intensity-laser therapy (HILT) group and ibuprofen gel phonophoresis (IGP) group. Duration of the treatment will be 8 minutes in one session/knee joint for each day for 3 days/week for 8 weeks.The pain and quality of life will be assessed at the baseline and at the end of 8-week post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with clinical knee OA according to the diagnostic criteria of ACR were included in the study

Exclusion Criteria:

* Unwillingness to participate in the study
* Recent history (within the last 3 months) of physical therapy to the same joint
* Recent history (within the last 3 months) of intra-articular procedure (injection and/or lavage) to the knee
* History of knee surgery/fracture
* Acute synovitis/arthritis including the infectious conditions
* Presence of malignancy
* Pregnancy
* Taking pain relief medications

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-05-21 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Digitalized pain pressure algometer (ALGO-DS-01) | Changes will be measured at baseline, end of 8-week post-intervention period
  Sensor digital algometer is force gauge with computer size which is highly accurate. The ALGO-DS-01 is chosen for the assessment of pain, which is a reliable and valid tool
Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC) | Changes will be measured at baseline, end of 8-week post-intervention period
  The Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC) will be used to evaluate the disease-specific self-reported symptoms of OA. This form is comprised of 24 questions in three categories including pain (5 questions), stiffness (2 questions), and physical function (17 questions).

SECONDARY OUTCOMES:
36-Item Short Form Health Survey (SF-36) | Changes will be measured at baseline, end of 8-week post-intervention period
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life (QoL). The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH).

CONTACTS AND LOCATIONS:
Overall Officials: Vipin Saini, Ph.D, Principal Investigator — Maharishi Markandeshwar Medical College and Hospital; Asir J Samuel, Principal Investigator — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation; Adarsh K Srivastav, MPT, Principal Investigator — Maharishi Markandeshwar Medical College and Hospital; Deeksha Sharma, MPT, Principal Investigator — Maharishi Markandeshwar Medical College and Hospital
Locations (1):
- Dr Vipin Saini, Solan, Himachal Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Larkin KA, Martin JS, Zeanah EH, True JM, Braith RW, Borsa PA. Limb blood flow after class 4 laser therapy. J Athl Train. 2012 Mar-Apr;47(2):178-83. doi: 10.4085/1062-6050-47.2.178. PMID 22488283
- [Result] de Matos Brunelli Braghin R, Libardi EC, Junqueira C, Rodrigues NC, Nogueira-Barbosa MH, Renno ACM, Carvalho de Abreu DC. The effect of low-level laser therapy and physical exercise on pain, stiffness, function, and spatiotemporal gait variables in subjects with bilateral knee osteoarthritis: a blind randomized clinical trial. Disabil Rehabil. 2019 Dec;41(26):3165-3172. doi: 10.1080/09638288.2018.1493160. Epub 2018 Oct 16. PMID 30324827
- [Result] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Result] Loyola-Sanchez A, Richardson J, Beattie KA, Otero-Fuentes C, Adachi JD, MacIntyre NJ. Effect of low-intensity pulsed ultrasound on the cartilage repair in people with mild to moderate knee osteoarthritis: a double-blinded, randomized, placebo-controlled pilot study. Arch Phys Med Rehabil. 2012 Jan;93(1):35-42. doi: 10.1016/j.apmr.2011.07.196. PMID 22200383
- [Result] Fransen M, McConnell S. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004376. doi: 10.1002/14651858.CD004376.pub2. PMID 18843657
- [Derived] Sharma D, Saini V, Srivastav AK, Samuel AJ. Comparative efficacy of high intensity laser therapy (Class IV) and ibuprofen gel phonophoresis in the treatment of knee osteoarthritis among people living in hilly terrain: A randomized controlled study. Lasers Med Sci. 2025 Oct 20;40(1):440. doi: 10.1007/s10103-025-04613-6. PMID 41114869